CLINICAL TRIAL: NCT06671834
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED, DOSE ESCALATION STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF MULTIPLE-DOSE TOPICAL ADMINISTRATION OF PF-07905428 IN HEALTHY PARTICIPANTS AND PARTICIPANTS WITH ACNE VULGARIS, AND ADDITIONALLY CLINICAL EFFECT IN PARTICIPANTS WITH MODERATE TO SEVERE ACNE VULGARIS AGED 18 TO 40 YEARS OLD
Brief Title: A Study to Learn About the Study Medicine Called PF-07905428 in Healthy Participants and Participants With Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C5441001; NCT06671834 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-10-18; First posted 2024-11-04 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- PF-07905428 Low Strength (Experimental): Participants may receive 0.08% PF-07905428 QD. Area of application will be increased as the study proceeds from one cohort to the next.
  Interventions: Drug: PF-07905428
- PF-07905428 High Strength (Experimental): Participants may receive 0.24% PF-07905428 QD. Area of application will be increased as the study proceeds from one cohort to the next.
  Interventions: Drug: PF-07905428
- Placebo (Placebo Comparator): All participants will receive Placebo QD. Area of application will be increased as the study proceeds from one cohort to the next.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-07905428 — Topical solution of PF-07905428 0.08% or PF-07905428 0.24%
  Arms: PF-07905428 High Strength; PF-07905428 Low Strength
Drug: Placebo — Topical solution of placebo
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to learn about the safety and effects of the study medicine (called PF-07905428) for the potential treatment of acne vulgaris.

This study is seeking participants who:

* Are male or female between the ages of 18 and 40
* Are generally healthy
* Are diagnosed with moderate to severe acne vulgaris (Cohort 4 only)

The study medicine will be applied every day on the participant's face and/or back for 14 days (Cohorts 1 and 2) or for 28 days (Cohort 3 and 4).

The investigators will compare the experiences of people receiving the study medicine to those of the people who do not. This will help the investigators determine if the study medicine is safe and effective.

Participants will take part in this study for approximately 2 months. During this time, they will have 17 study visits (Cohorts 1 and 2) or 31 study visits (Cohorts 3 and 4) at the study clinic. The study team will also call participants once at the end of the study over the phone.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation.
* Only for participants who are enrolling with acne vulgaris: diagnosis of acne vulgaris for 3 months or greater
* For participants enrolling in Cohort 1-3 with acne vulgaris (optional): mild to moderate facial acne vulgaris
* For participants enrolling in Cohort 4 with acne vulgaris: moderate to severe facial acne vulgaris

Exclusion Criteria:

* Participants with very severe acne
* Participants with autoinflammatory syndromes
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C.
* Participants with clinically significant laboratory abnormalities

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-12-04 (Actual); Study Completion 2025-12-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Through study completion, approximately 2 months
  An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were events between first dose of study drug and up to 37 days after last dose that were absent before treatment or that worsened relative to pretreatment state. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs included SAEs and all non-SAEs that occurred during the study.
Number of Participants With Clinical Laboratory Abnormalities | Through study completion, approximately 2 months
  Evaluation of participants with clinically meaningful changes from baseline in laboratory test results
Number of Participants With Abnormalities in Vital Signs | Through study completion, approximately 2 months
  Any untoward vital sign findings that are identified during the active collection period and meet the definition of an AE or SAE.
Number of Participants With Clinically Significant Changes From Baseline in 12-Lead Electrocardiogram (ECG) Parameters | Through study completion, approximately 2 months
  12-lead ECG were performed after the participant had rested quietly for at least 10 minutes in a supine position. ECG parameters included RR interval, PR interval, QRS complex, QT interval, corrected QT (QTc) interval, Bazett's correction QT (QTcB) interval, Heart Rate and Fridericia's correction (QTcF) interval. Clinical significance of 12-Lead ECG was judged by investigator.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of PF-07905428 | Day 14 (Cohorts 1, 2, and 4) Day 28 (Cohorts 3 and 4)
Time to maximum plasma concentration (Tmax) of PF-07905428 | Day 14 (Cohorts 1, 2, and 4) Day 28 (Cohorts 3 and 4)
Area Under the Serum Concentration-Time Curve Over the Dosing Interval (AUCtau) of PF-07905428 | Day 14 (Cohorts 1, 2, and 4) Day 28 (Cohorts 3 and 4)
  Area under the plasma concentration-time curve from time 0 to the end of the dosing interval (AUCtau)
Terminal serum elimination half life (t1/2) of PF-07905428 | Day 14 (Cohorts 1, 2, and 4) Day 28 (Cohorts 3 and 4)
Absolute change in total acne lesion counts | Baseline to Week 4
  To compare the clinical effect of PF-07905428 versus placebo on absolute change from baseline in total lesion count (TLC) in participants with moderate to severe acne vulgaris.
Absolute change from baseline in inflammatory lesion counts (ILC) | Baseline to Week 4
  To compare the clinical effect of PF-07905428 versus placebo on absolute change from baseline in inflammatory lesion counts (ILC) in participants with moderate to severe acne vulgaris.
Absolute change in non-inflammatory lesion counts (nILC) | Baseline to Week 4
  To compare the clinical effect of PF-07905428 versus placebo on absolute change from baseline in non-inflammatory lesion counts (nILC) in participants with moderate to severe acne vulgaris.
Percentage of Participants who achieve Investigator global assessment (IGA) of 0 or 1 | Baseline to Week 4
  Percentage of participants who achieve IGA score of "clear" or "almost clear" on the face (modified IGA of 0 or 1) with 2-points or greater improvement at Week 4 compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Innovaderm Research Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5441001